CLINICAL TRIAL: NCT04883645
Title: Pilot Clinical Trial of Neoadjuvant Toll-like Receptor 7 Agonist (Imiquimod) Immunotherapy in Early-Stage Oral Squamous Cell Carcinoma
Brief Title: Neoadjuvant Imiquimod Immunotherapy for Oral Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103625; 7R21CA252441-02 (NIH)
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Topical Aldara (Experimental): All patients receive the same treatment (there is no "placebo" arm). Treatment will be self-administered by the patients on an outpatient basis. All patients with untreated and biopsy confirmed oral squamous cell carcinoma (OSCC) who meet the inclusion criteria.
  Interventions: Drug: Imiquimod 5% Cream

INTERVENTIONS:
Drug: Imiquimod 5% Cream — Imiquimod as a 5% cream is being used to treat several skin cancers, including malignant melanoma, basal cell carcinoma (BCC) and SCC. With respect to SCC treatment, it has been demonstrated that imiquimod stimulates tumor destruction by recruiting T cells (cells in the immune system) from blood and by inhibiting tonic anti-inflammatory signals within the tumor. The patient will be instructed to apply imiquimod cream, 7 nights a week for 4 weeks to the oral tumor at bedtime.
  Other Names: Aldera

SUMMARY:
The purpose of this research study is to find out what effects, good and/or bad, topical application of the drug Aldara will have on patients and on their oral cancer. Aldara is a drug that activates toll-like receptor (TLR) in oral cancer cells causing self-destruction of tumor cells. It also activates immune cells to attack and eliminate cancer cells. Aldara is currently approved by the Food and Drug Administration (FDA) for treatment of skin cancer and melanoma. Its use in this study is 'off-label' (use of a drug approved by FDA for skin cancer to treat oral cancer in this study).

The preliminary efficacy of topical imiquimod in a neoadjuvant setting in patients with early-stage oral squamous cell carcinoma will be determined by a reduction in tumor cellularity in post-treatment tissue compared to pre-treatment tissue. Safety and tolerability will be evaluated by CTCAE v5 criteria. The effect of imiquimod on the tumor immune microenvironment will be assessed by performing quantitative multiplex immunofluorescence.

DETAILED DESCRIPTION:
The researchers propose an exploratory clinical trial to evaluate the efficacy of topical imiquimod, a TLR-7 agonist, in patients with early-stage oral squamous cell carcinoma. The analysis of pre- and post-treatment tumor specimen collected from patients treated on this study will be used for quantitative immunoflourescence analysis to assess the immunomodulatory activity of imiquimod in human tumor samples. The researchers hypothesize that TLR-7 stimulation will reduce the size of the tumor in patients with early-stage oral squamous cell carcinoma. The researchers anticipate that activation of immune cells will correlate with response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated and biopsy confirmed oral squamous cell carcinoma (OSCC)
* Clinical (TNM) stage I or II
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2

Exclusion Criteria:

* Patients associated with prior therapy requiring treatment with systemic immunosuppressive treatments with the exception of vitiligo, childhood asthma that has resolved, residual endocrinopathies requiring replacement therapy, or psoriasis that does not require systemic treatment
* Treatment with any other investigational agents
* Requirement for immunosuppressive intraoral topical or systemic corticosteroids prior to the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV positive patients on combination antiretroviral therapy
* Have evidence of any other significant oral mucosal condition, clinical disorder, physical examination finding, or laboratory finding that, as judged by the investigator, makes it undesirable for the patient to participate in the study
* Pregnant women are excluded from this study because imiquimod may have adverse effect on the fetus (FDA pregnancy risk category C). Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with imiquimod, breastfeeding should be discontinued if the mother is receiving study treatment
* Male patients unwilling or unable to comply with pregnancy prevention measures
* Subjects not receiving initial surgical treatment at Medical University of South Carolina (MUSC)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Yoon, DDS, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon AJ, Carvajal RD, Graboyes EM, Kaczmar JM, Albergotti WG, Kejner AE, Troob SH, Philipone E, Anoma JS, Armeson KE, Hill EG, Richardson MS, Woods TR, Chera BS, Nourollah-Zadeh F, Lee BJ, Pandruvada S, Kourtidis A, Kingsley C, O'Quinn EC, Mills S, Jordan VC, Spencer M, Fails D, McKee TD, Zaidi M, Brisendine A, Horn S, Mehrotra S, Ogretmen B, Newman JG. Pilot clinical trial of neoadjuvant toll-like receptor 7 agonist (Imiquimod) immunotherapy in early-stage oral squamous cell carcinoma. Front Immunol. 2025 Jan 27;16:1530262. doi: 10.3389/fimmu.2025.1530262. eCollection 2025. PMID 39931064

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: Topical Aldara
Started | 16
Completed | 15
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Early-stage oral squamous cell carcinoma
Groups:
- Imiquimod Treatment: All patients receive the same treatment (there is no "placebo" arm). Treatment will be self-administered by the patients on an outpatient basis. All patients with untreated and biopsy confirmed oral squamous cell carcinoma (OSCC) who meet the inclusion criteria.
  Imiquimod 5% Cream: Imiquimod as a 5% cream is being used to treat several skin cancers, including malignant melanoma, basal cell carcinoma (BCC) and SCC. With respect to SCC treatment, it has been demonstrated that imiquimod stimulates tumor destruction by recruiting T cells (cells in the immune system) from blood and by inhibiting tonic anti-inflammatory signals within the tumor. The patient will be instructed to apply imiquimod cream, 7 nights a week for 4 weeks to the oral tumor at bedtime.
Arm/Group | Imiquimod Treatment
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: Years] | 65 [52 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 50% Reduction in Tumor Cell Count and Major Pathologic Response
Description: A minimum of 50% reduction in tumor cell count assessed by quantitative multiplex immunofluorescence (qmIF) within the tumor bed of the surgical tissue (post-treatment) compared to the biopsy tissue (pre-treatment). In addition, the major pathologic response to be assessed using Immune-Related Pathologic Response Criteria (irPCR) in the tumor bed of the post-treatment surgical tissue.
Time Frame: Following 28 days of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Imiquimod: All patients receive the same treatment (there is no "placebo" arm). Treatment will be self-administered by the patients on an outpatient basis. All patients with untreated and biopsy confirmed oral squamous cell carcinoma (OSCC) who meet the inclusion criteria.
  Imiquimod 5% Cream: Imiquimod as a 5% cream is being used to treat several skin cancers, including malignant melanoma, basal cell carcinoma (BCC) and SCC. With respect to SCC treatment, it has been demonstrated that imiquimod stimulates tumor destruction by recruiting T cells (cells in the immune system) from blood and by inhibiting tonic anti-inflammatory signals within the tumor. The patient will be instructed to apply imiquimod cream, 7 nights a week for 4 weeks to the oral tumor at bedtime.
Arm/Group | Experimental: Imiquimod
Number analyzed (Participants) | 15
Participants
  Greater than 50% reduction and Major Pathologic Response | 9
  Less than 50% reduction and Partial Response | 6

2. Secondary Outcome: Safety of Imiquimod Therapy
Description: Defined as safe no life-threatening (Grade 4) adverse events assessed by CTCAE v5 criteria.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Imiquimod
Number analyzed (Participants) | 15
Participants
  Grade 4 AEs | 0
  No Grade 4 AEs | 15

3. Other Pre Specified Outcome: Changes in Immune Cell Count
Description: To assess the changes in anti-tumoral immune cell counts from pre- to post-therapy by quantitative multiplex immunofluorescence (normalized cell number per mm^2 from 6 to 8 regions of interest).
Time Frame: Following 28 days of treatment
Measure: Median (95% Confidence Interval); unit: Normalized cells/mm^2
Groups:
- Correlative: Change in Antitumor Immune Cell Count After Imiquimod Immunotherapy.: All patients receive the same treatment (there is no "placebo" arm). Treatment will be self-administered by the patients on an outpatient basis. All patients with untreated and biopsy confirmed oral squamous cell carcinoma (OSCC) who meet the inclusion criteria.
Arm/Group | Correlative: Change in Antitumor Immune Cell Count After Imiquimod Immunotherapy.
Number analyzed (Participants) | 15
Normalized cells/mm^2
  Contribution of Increase in Functional Helper T cells in Reduction in Tumor | 0.54 [0.06 to 0.84]
  Contribution of Increase in Activated Cytotoxic T cells in Tumor Reduction | 0.55 [-0.06 to 0.97]

4. Other Pre Specified Outcome: RFS Follow-up
Description: One-year relapse-free survival (RFS)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Correlative: Shift in Antitumor Immune Profile After Imiquimod Immunotherapy.: All patients receive the same treatment (there is no "placebo" arm). Treatment will be self-administered by the patients on an outpatient basis. All patients with untreated and biopsy confirmed oral squamous cell carcinoma (OSCC) who meet the inclusion criteria.
Arm/Group | Correlative: Shift in Antitumor Immune Profile After Imiquimod Immunotherapy.
Number analyzed (Participants) | 14
Participants
  One-year RFS | 13
  Recurrence within one-year | 1

ADVERSE EVENTS:
Time Frame: Two months
Description: The secondary endpoint was treatment-related toxicity graded by CTCAE v5, defined as safe if no life-threatening (Grade 4) is reported.
Groups:
- Imiquimod: Treatment group
Arm/Group | Imiquimod
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imiquimod (N=16)
Mortality (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imiquimod (N=16)
Oral mucositis (Investigations) | 14 (14)
Oral pain/Sore throat (Investigations) | 6 (6)
Fatigue (Investigations) | 2 (2)
Oral hemorrhage (Investigations) | 1 (1)
Nausea (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT04883645/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT04883645/ICF_000.pdf